CLINICAL TRIAL: NCT02048111
Title: Pharmacokinetics, Safety and Efficacy of Recombinant Factor IX Product, IB1001, in Patients With Severe Hemophilia B
Brief Title: Study of Recombinant Factor IX Product, IB1001, in Previously Treated Subjects With Hemophilia B
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn from the IND.
Sponsor: Cangene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IB1001-04
Record Dates: First submitted 2013-11-14; First posted 2014-01-29 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Hemophilia A; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked
MeSH Terms: conditions — Hemophilia B; Hemophilia A; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked | interventions — IB1001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IB1001 (Experimental)
  Interventions: Biological: IB1001

INTERVENTIONS:
Biological: IB1001 — Prophylaxis (during Treatment and Continuation phases): 40 - 75 IU/kg twice weekly.
  The starting dose for prophylaxis may be based on previous recombinant factor IX product use. The recommended starting prophylaxis dose is 40 - 60 IU/kg twice weekly, however, the investigator may prescribe up to 75 IU/kg twice weekly at their discretion (after clinically assessing the subject) and discretion of the subject.
  The dose or the frequency of IB1001 prophylaxis may be adjusted at the discretion of the investigator.

SUMMARY:
To evaluate the safety (acute adverse effects associated with infusions, and inhibitor development), pharmacokinetics (PK), and efficacy with respect to breakthrough bleeding and control of hemorrhaging during prophylaxis of IB1001 in subjects with hemophilia B.

DETAILED DESCRIPTION:
Primary Objectives:

* to evaluate safety of IB1001 within the first 50 exposure days,
* to determine IB1001 pharmacokinetics (PK), and
* to assess efficacy of IB1001 prophylaxis with respect to breakthrough bleeding and with respect to control of hemorrhaging in subjects with severe hemophilia B within the first 50 exposure days

Secondary Objectives:

* to evaluate long-term safety of IB1001; and
* to evaluate long term efficacy of IB1001.

Exploratory Objectives:

* to evaluate markers of thrombogenicity during the first 24 hours post-infusion [thrombogenicity markers will include at a minimum D-dimer test; however should there be a clinical reason (e.g., three consecutive elevations in D-dimer levels, a possible clinical thrombogenic episode), sufficient samples will be collected to also evaluate levels of fragment 1+2 (F1+2) and thrombin-antithrombin III complex (TAT)]
* to evaluate IB1001 immunogenicity response (development of inhibitory and non-inhibitory factor IX binding antibodies and antibodies to host cell proteins)

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 12 years
2. Body Mass Index of ≤ 29, with a minimum body weight of 40 kg
3. Written Institutional Review Board (IRB)/ Ethics Committee (EC)-approved informed consent form (ICF)
4. Willingness to make the required study visits, and follow instructions while enrolled in the study (up to 12 months)
5. Severe (factor IX activity ≤2 U/dL) hemophilia B patients with a minimum of 3 bleeding episodes over the preceding 6 months or 6 bleeding episodes over the preceding 12 months or in the event the subject is on prophylaxis, a minimum of 3 bleeding episodes over the preceding 6 months or 6 bleeding episodes over the preceding 12 months prior to being placed on prophylaxis
6. Subjects must be on prophylaxis or switch to a prophylaxis regimen for the duration of the PK and Treatment/Continuation Phase of the study
7. Previously treated patients with a minimum of 150 exposure days to a factor IX preparation
8. Willingness to adhere to the 5-day washout of any factor IX replacement therapy prior to PK evaluations
9. Immunocompetent (CD4 count >400/mm3) and not receiving immune modulating or chemotherapeutic agents
10. Platelet count at least 150,000/mm3
11. Liver function: alanine transaminase (ALT) and aspartate transaminase (AST) ≤2 times the upper limit of the normal range
12. Total bilirubin ≤1.5 times the upper limit of the normal range
13. Renal function: serum creatinine ≤1.25 times the upper limit of the normal range
14. Hemoglobin ≥7 g/dL at the time of the blood draw

Exclusion Criteria:

1. History of factor IX inhibitor ≥0.6 BU (Bethesda units)
2. Existence of another coagulation disorder
3. Evidence of thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC)
4. Use of an investigational drug within 30 days prior to study entry
5. Previous use of IB1001
6. Use of medications that could impact hemostasis, such as aspirin
7. Hypersensitivity to the active substance or to any of the excipients in the investigational products
8. Known allergic reaction to hamster proteins
9. History of poor compliance, a serious medical or social condition, or any other circumstance that, in the opinion of the investigator, would interfere with participation or compliance with the study protocol
10. History of adverse reaction to either plasma-derived factor IX or recombinant factor IX that interfered with the subject's ability to treat bleeding episodes with a factor IX product

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of study subjects with adverse events | Within 6 months
  Information on adverse events is collected after each infusion of study drug by a study subject. Assessment of adverse events is then performed by an investigator after 5 infusions of study drug, 1 month, 2 months, 3 months and 6 months of study drug treatment.

SECONDARY OUTCOMES:
Number of bleeding episodes divided by number of months of observation | Within 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Chicago, Illinois, United States
- Manchester, United Kingdom